CLINICAL TRIAL: NCT01824368
Title: FOTOAFERESIS EXTRACORPÓREA EN EL TRASPLANTE HEPÁTICO. ENSAYO CLINICO EN FASE II DE SEGURIDAD Y EFICACIA EN PACIENTES CON RETIRADA PROGRESIVA DE LA INMUNOSUPRESIÓN
Brief Title: Extracorporeal Photopheresis in Liver Transplantation. Phase II Clinical Trial in Safety and Efficacy in Patients With Gradual Decrease of Immunosuppression.
Acronym: FEC-TH
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Red de Terapia Celular (Industry)
Collaborators: Spanish National Health System (Other); Universidad de Murcia (Other); Hospital Universitario Virgen de la Arrixaca (Other); Public Health Service, Murcia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FEC-TH; 2012-000633-39 (EudraCT Number)
Record Dates: First submitted 2013-04-01; First posted 2013-04-04 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2016-04

CONDITIONS: Liver Transplantation; Immunosuppression
MeSH Terms: interventions — FEC protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- People with liver transplantation (Experimental): People with liver transplantation over 2 years following treatment with immunosuppression including cyclosporine or tacrolimus.
  Interventions: Procedure: Extracorporeal Photopheresis Procedure (FEC)

INTERVENTIONS:
Procedure: Extracorporeal Photopheresis Procedure (FEC) — The FEC will be held in the Cellex (Therakos), and authorized device in routine use in our unit for performing FEC in the treatment of graft-versus-host and cutaneous T-cell lymphoma. After performing a blood count, will connect the patient to Cellex through a central or peripheral.
  1500 mL typically be processed peripheral blood mononuclear fraction obtained by apheresis process. Then be added Uvadex (8-metoxipsolareno, 0.017 mL / mL) to the mononuclear fraction bag and proceed to photoactivation with UVA radiation.
  Finally the photoactivated product is again infuse the patient. It will monitor the final blood count to assess hemoglobin and platelets. The entire procedure is performed in a single step and closed mode, with Cellex.

SUMMARY:
The purpose of this study is to evaluate the safety of extracorporeal photopheresis in patients with long-standing liver transplantation subjected to a progressive reduction of immunosuppression by complications arising from its use.

ELIGIBILITY:
Inclusion Criteria:

* Have been receiving liver transplant two years ago.
* Be 18 years or older.
* Treatment with immunosuppression including cyclosporine or tacrolimus.
* Having a normal liver function in the last year
* Not have suffered acute rejection in the last year and have no chronic rejection
* Submit any significant side effects from medication immunosuppressive (hypertension, creatinine greater than 1.7 mgDl, diabetes, morbid obesity, osteoporosis, hyperlipidemia, severe hirsutism, neurotoxicity novo malignancy, etc.)
* Etiology of underlying disease: alcoholic cirrhosis with or without hepatocarcinoma, metabolic diseases, amyloidotic polyneuropathy family, biliary atresia, fulminant hepatitis non-A, non-B, non-C, cirrhosis cryptogenic and generally causes no viral or autoimmune.
* Patients offering sufficient guarantees of adherence to protocol
* Patients who give written informed consent for participate in the study.
* It is necessary that the patient meets all inclusion criteria.

Exclusion Criteria:

* Underlying disease of the autoimmune (primary sclerosing cholangitis, autoimmune cirrhosis, primary biliary cirrhosis) or epatocarcinoma about cirrhosis of viral or autoimmune.
* Patients with chronic rejection, or acute rejection in the last year.
* Patients with liver retransplantation.
* patients with history of hypersensitivity or idiosyncratic reactions to methoxsalen, psoralen the compounds or any of the excipients.
* patients with melanoma, cutaneous basal cell carcinoma or squamous cell coexistent.
* Patients with aphakia.
* Patients taking Oxoralen.
* Pregnant women or nursing mothers, or adults of childbearing age not using effective contraception.
* Participation in another clinical trial.
* Inability to understand informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
adverse event rate and rate of transplant rejection | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Virgen de la Arrixaca, El Palmar, Murcia, Spain

REFERENCES:
- See also: Red de Terapia Celular (TerCel) — http://www.red-tercel.com
- See also: Fundación para la Formación e Investigación Sanitarias Región de Murcia — http://www.ffis.es
- See also: Servicio Murciano de Salud — http://www.murciasalud.es